CLINICAL TRIAL: NCT00262665
Title: Randomized, Placebo-controlled Trial of an AMPAkine in Major Depressive Disorder
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: protocol cancelled
Sponsor: Dennis Charney (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor-Investigator, Dennis Charney, Dean, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GCO # 05-0384
Record Dates: First submitted 2005-12-06; First posted 2005-12-07 (Estimated); Last update posted 2012-12-11 (Estimated); Status verified 2012-12

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — 1-(benzofurazan-5-ylcarbonyl)piperidine; AMPA receptor potentiator HBT1

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Org 24448 (Experimental): ampa receptor potentiator for the treatment of MDD
  Interventions: Drug: ORG 24448
- Placebo (Placebo Comparator): matching placebo pill
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ORG 24448 — flexible regimen starting at 250mg once a day, increasing to maximum of 750mg twice a day.
  Other Names: AMPA receptor potentiator
  Arms: Org 24448
Drug: Placebo — matching placebo pill - flexible regimen starting at 250mg once a day, increasing to maximum of 750mg twice a day.
  Arms: Placebo

SUMMARY:
The purpose of this study is to test a candidate drug, Org 24448,in a phase II clinical trial in adult patients with moderately treatment-resistant unipolar major depressive disorder.

DETAILED DESCRIPTION:
Major depressive disorder (MDD) is a common, severe, chronic and often life-threatening illness. Major depression contributes to significant morbidity and mortality. Available pharmacotherapies for major depression are suboptimal in terms of speed of onset, efficacy, and tolerability. Current medications for severe, chronic mood disorders are not based on pathophysiological models of illness, but rather are variation of monoaminergic-based therapies. Org 24448 represents a new treatment approach for depression, by potentiating the AMPA receptor subfamily of ionotropic glutamate receptors. This drug has been shown to have antidepressant features in preclinical models, as well as cognitive-enhancing qualities.

ELIGIBILITY:
Inclusion Criteria:

* Clinical Diagnosis of MDD
* Have not responded to an adequate trial of one antidepressant in the current episode or have not completed antidepressant trials due to intolerance to ≤3 antidepressant medications in the current or a previous episode

Exclusion Criteria:

* Presence of psychotic features, OCD, drug or alcohol dependency with the preceding 3 months

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2005-03; Primary Completion 2005-03 (Actual); Study Completion 2005-03 (Actual)

PRIMARY OUTCOMES:
mean change in the Montgomery-Asberg Depression Rating Scale (MADRS) from baseline to 8 weeks | at baseline and at 8 weeks
  Reduction of depressive symptoms as measured by the Montgomery-Asberg Depression Rating Scale (MADRS) at 8 weeks as compared to baseline.

SECONDARY OUTCOMES:
change in neuropsychological function from baseline to 7 weeks | at baseline and at 7 weeks
  Effect on neuropsychological functioning measured by neuropsychological testing

CONTACTS AND LOCATIONS:
Overall Officials: Dennis S Charney, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai